CLINICAL TRIAL: NCT04868305
Title: Randomized Clinical Trial: Treatment of Unstable Trochanteric Hip Fractures With Intramedullary Nail Versus Hip Arthroplasty: Survival, Complications and Postoperative Patient Reported Outcomes
Brief Title: Intramedullary Nail Versus Hip Arthroplasty in Unstable Trochanteric Hip Fractures
Acronym: TUFHIPRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140120V1
Record Dates: First submitted 2021-04-06; First posted 2021-04-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-11

CONDITIONS: Hip Injuries and Disorders; Hip Fractures
Keywords: Trochanteric hip fracture; Unstable trochanteric hip fractures
MeSH Terms: conditions — Hip Injuries; Disease; Hip Fractures | interventions — Fracture Fixation, Intramedullary; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Patients with an identified unstable trochanteric hip fracture (AO 31A2.2-3.3) who has fulfilled inclusion criteria and given their consent will be randomized into one of two treatments; Intramedullary nail versus hip arthroplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramedullary nail (Active Comparator): Intramedullary nail with proximal lagscrew and distal locking screw(s)
  Interventions: Procedure: Intramedullary nail
- Hip arthroplasty (Active Comparator): Hemiarthroplasty (HA) or Total hip arthroplasty (THA). A cemented dual-mobility cup will be utilized in THA. Addition of cerclage/trochanter claw plate to fixate trochanter major will be used when suitable.
  Interventions: Procedure: Hip arthroplasty

INTERVENTIONS:
Procedure: Intramedullary nail — Intertan nail (Smith & Nephew)* or Gamma 3 nail (Stryker)*
  * All of the above-mentioned products are subjects to change into an equivalent product
  Arms: Intramedullary nail
Procedure: Hip arthroplasty — Total hip arthroplasty:
  * Cemented: Lubinus (Link)*, Exeter (Stryker)*
  * Uncemented: Restoration Modular (Stryker)*
  * Cup: Cemented Avantage dual mobility cup (Zimmer Biomet)*
  Hemiarthroplasty:
  * Cemented: Lubinus (Link)*, Exeter (Stryker)*
  * Uncemented: Restoration Modular (Stryker)*
    * All of the above-mentioned products are subjects to change into an equivalent product
  Arms: Hip arthroplasty

SUMMARY:
A hip fracture is a large burden to the patient with increased mortality, pain and increased need for daily assistance. Trochanteric fractures of the femur (FTF) represents about 35% of the hip fractures. Today FTFs are mainly treated with internal fixation using sliding hips screws (SHS) or intramedullary nail (IMN), whilst hip arthroplasty (THA/HA) is rarely used. Despite advances in the design of the internal fixation implants there is a high failure rate, in particular in cases of FTFs classified as unstable fractures. Since the introduction of hip arthroplasty in femoral neck fractures there has been a reduction in complication rates, early mobilization and shorter hospital stays.

The primary objective of this project is to investigate if treatment with hip arthroplasty in unstable FTFs will increase the postoperative mobility, give a better general health outcome for the patient, better quality of life and reduce re-operation rate for the patients compared to those operated with the traditional IMN.

DETAILED DESCRIPTION:
Proximal femoral fractures also termed "hip" fractures are one of the most common fractures among adults over 50 years of age. With increase in life expectancy, the incidence of these fractures is also increasing. By 2040, the number of these fractures are expected to double in Norway. Trochanteric fractures of the femur (Fractura Trochanterica Femoris, FTF) represents about 35% of the hip fractures in Norway . There are many classification systems for FTFs, but The Orthopaedic Trauma Association (OTA) have adopted the system developed by the Arbeitsgemeinschaft Osteosynthese (AO ) group, and is the most commonly used in addition to the Evans Jensens classification.

The mean age of hip fracture patients is 82 years for women and 78 for men. The comorbidity in this patient group is high with large amount of dementia, sarcopenia and osteoporosis. The one-year mortality rate after a hip fractures is 20-35%. According to the Norwegian Hip Fracture Register 15 % of the hip fractures are unstable trochanteric fractures (AO 31A2.2-A3). The prognosis is poor, in particular for unstable (multi fragmented) fractures, with reported complications up to 35-51 %.

Substantial research has established better understanding and best practice guidelines to treat the femoral neck fractures, mostly with hip arthroplasty, however no superior method is established for the unstable trochanteric fractures. 'Getting It Right First Time' is important for these fragile patients, thus post-operative complications are associated with a large increase in the mortality.

Today, most of the FTFs are reduced and fixated with a sliding hip screw (SHS), although the use of intramedullary nails (IMN) is increasing. RCTs have shown better survival of IMN compared to SHS for the more distal FTFs and subtrochanteric fracture. Unstable FTFs (AO 31A2 - A3, EVJ III-V) have high reoperation rates (21-35%) when operated either with SHS or IMN. Unacceptable shortening, external rotation deformity of the limb and long time to recover/mobilization have been the problems with osteosynthesis.

The question is if hip arthroplasty can give a superior treatment outcome for patients suffering from unstable subtypes of trochanteric hip fractures compared to the traditional treatment with IMN. A randomized clinical trial is to be conducted comparing these two treatment methodologies.

Stavanger University Hospital (SUH) receives over 150 FTFs per year. About 1/3 of the FTFs are of unstable fracture morphology. The planned study is a randomized clinical trial. The randomization module will be provided by Klinisk forskningsenhet Midt-Norge (KlinForsk). Patients fulfilling the inclusion criteria will be randomized to one of two treatment groups, IMN versus hip arthroplasty.

Included patients will be treated in accordance to a local operation protocol:

Intramedullary nails will be operated by a resident orthopedic surgeon with at least 2 years' experience in fracture surgery or a consultant orthopedic surgeon (there must always be a consultant orthopedic surgeon present in the surgical team). A long IMN must always be utilized. Anatomical reposition or positive anterior and medial cortical support should be strived to be achieved. If a large antero- or posteromedial fragment is present one should consider an additional cerclage to fix the fragment.

Arthroplasty will be operated by a resident orthopedic surgeon with at least 2 years' experience with hip arthroplasty surgery or by a consultant orthopedic surgeon subspecialized in arthroplasty surgery, with competency within revision or difficult primary hip arthroplasty surgery (there must always be a consultant orthopedic surgeon subspecialized in arthroplasty surgery present in the surgical team). Posterior surgical approach will be used. If a cup is to be utilized it must be a cemented dual-mobility cup.

The patients will have follow-up appointments at 2-, 6 and 12 months postoperative. Following data will be collected:

* Patient reported outcome measures (HOOS and EQ5D)
* Timed up and go test
* Trendelenburg test
* Clinical leg length discrepancy
* Radiological assessment from hip x-rays (AP and lateral)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* American Society of Anesthesiology Score (ASA) < 4
* Ambulant with or without aid (preinjury)
* Radiological verified unstable trochanteric hip fracture (AO 31A2.2 - 3.3)
* Written consent obtained by patient or his/her next of kin

Exclusion Criteria:

* Previous hip surgery on ipsilateral or contralateral side
* Non-ambulant preinjury
* Patient not living in the area of hospital care

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome Measure (PROM) | Collected at 2, 6 and 12 months from primary surgery
  Hip disability and Osteoarthritis Outcome Score (HOOS).
  "HOOS is developed as an instrument to assess the patients' opinion about their hip and associated problems. HOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related Quality of life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The result can be plotted as an outcome profile.
  * Above information about HOOS is copied from the authors of www.KOOS.nu
  * Change in HOOS score will be observed from 2-, 6- and 12 months.
Patient Reported Outcome Measure (PROM) | Collected from 2 to 12 months from primary surgery
  EuroQol EQ-5D.
  "The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement."
  Change in EQ-5D score will be observed from 2-, 6- and 12 months.

SECONDARY OUTCOMES:
Mortality | 2, 6 and 12 months from primary surgery
  Mortality rates will be analyzed
Complications related to prosthesis | Collected from 2 to 12 months from primary surgery
  Specific complications related to the randomly assign intervention;
  * Peri prosthesis fracture
  * Prosthesis dislocation
  * Prosthesis loosening
  * Dislocation of trochanter major
  * Surgical wound infection (superficial)
  * Deep surgical wound infection
Complications related to osteosynthesis | Collected from 2 to 12 months from primary surgery
  Specific complications related to the randomly assign intervention;
  * Peri implant fracture (intraoperative or postoperative)
  * Implant cut-out
  * Non-union of fracture
  * Dislocation of trochanter major
  * Surgical wound infection (superficial)
  * Deep surgical wound infection
Somatic postoperative complications | Collected from 2 to 12 months from primary surgery
  * Deep vein thrombosis or other thromboembolic event
  * Pressure sores
  * Neurological complications
  * Other
Reoperation rate | Collected at 2, 6 and 12 months from primary surgery
  Reoperation rate (and causes) within each intervention arm
Radiological assessment of horizontal center of rotation (prosthesis) | Collected at 2, 6 and 12 months from primary surgery
  Horizontal center of rotation (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of vertical center of rotation (prosthesis) | Collected at 2, 6 and 12 months from primary surgery
  Vertical center of rotation (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of acetabular inclination (prosthesis) | Collected at 2, 6 and 12 months from primary surgery
  Acetabular inclination (degrees)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of acetabular anteversion (prosthesis) | Collected at 2, 6 and 12 months from primary surgery
  Acetabular anteversion (degrees)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of femoral stem positioning (prosthesis) | Collected at 2, 6 and 12 months from primary surgery
  Femoral stem positioning (valgus, neutral, varus)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of leg length discrepancy (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Leg length discrepancy (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of femoral neck length (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Femoral neck length (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of hip offset (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Hip offset (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of tip-to-apex (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Tip-to-Apex (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of medial cortical support (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Medial cortical support (negativ, neutral or positive)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of anterior cortical support (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Anterior cortical support (negativ, neutral or positive)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Radiological assessment of trochanter major dislocation (intramedullary nail) | Collected at 2, 6 and 12 months from primary surgery
  Trochanter major dislocation (millimeter)
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Timed Up and Go test (TUG test) | Collected at 2, 6 and 12 months from primary surgery
  Timed Up and Go test is used to asses mobility at follow-up 2-, 6- and 12 months postoperative.
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.
Trendelenburg test | Collected at 2, 6 and 12 months from primary surgery
  Trendelenburg test is used to assess hip abductor function at follow-up 2-, 6- and 12 months postoperative.
Clinical leg length discrepancy | Collected at 2, 6 and 12 months from primary surgery
  Clinical assessment of leg length discrepancy using 5 mm plates.
  Observation for eventual changes in above mentioned variable will be recorded throughout three follow-up appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Ane Djuv, MD., PhD, Principal Investigator — Helse Stavanger HF; Jan-Erik Gjertsen, MD., PhD, Study Chair — Haukeland University Hospital
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No